CLINICAL TRIAL: NCT01763905
Title: A Double-blind, Randomized, Multicenter Study to Evaluate Safety and Efficacy of AMG 145, Compared With Ezetimibe, in Hypercholesterolemic Subjects Unable to Tolerate an Effective Dose of a HMG-CoA Reductase Inhibitor
Brief Title: Goal Achievement After Utilizing an Anti-PCSK9 Antibody in Statin Intolerant Subjects -2
Acronym: GAUSS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110116; 2012-001364-30 (EudraCT Number)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Hyperlipidemia
Keywords: High Cholesterol, Treatment for high cholesterol, Lowering cholesterol, Lowering high cholesterol, Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — evolocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ezetimibe (Q2W) (Active Comparator): Participants received placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe orally once a day for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Ezetimibe
- Ezetimibe (QM) (Active Comparator): Participants received placebo subcutaneous injection once a month and 10 mg ezetimibe orally once a day for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Ezetimibe
- Evolocumab Q2W (Experimental): Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Placebo to Ezetimibe
- Evolocumab QM (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Placebo to Ezetimibe

INTERVENTIONS:
Biological: Evolocumab — Subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab Q2W; Evolocumab QM
Drug: Placebo to Evolocumab — Subcutaneous injection
  Arms: Ezetimibe (Q2W); Ezetimibe (QM)
Drug: Ezetimibe — Tablet for oral administration
  Other Names: Zetia
  Arms: Ezetimibe (Q2W); Ezetimibe (QM)
Drug: Placebo to Ezetimibe — Tablet for oral administration
  Arms: Evolocumab Q2W; Evolocumab QM

SUMMARY:
The primary objective was to evaluate the effect of 12 weeks of subcutaneous (SC) evolocumab every 2 weeks (Q2W) and monthly (QM), compared with ezetimibe, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in hypercholesterolemic adults unable to tolerate an effective dose of a statin (HMG-CoA (5-hydroxy-3-methylglutaryl-coenzyme A) reductase inhibitors).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 80 years of age
* Not on a statin or on a low dose statin with stable dose for at least 4 weeks
* History of intolerance to at least 2 statins
* Subject not at LDL-C goal
* Lipid lowering therapy has been stable prior to enrolment for at least 4 weeks.
* Fasting triglycerides ≤ 400 mg/dL

Exclusion Criteria:

* New York Heart Association (NYHA) III or IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Type 1 diabetes, poorly controlled type 2 diabetes
* Uncontrolled hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2013-11-19 (Actual); Study Completion 2013-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (56):
- United States (18):
  - Research Site, Carmichael, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Thousand Oaks, California
  - Research Site, Atlanta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Auburn, Maine
  - Research Site, Traverse City, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Houston, Texas
- Australia (4):
  - Research Site, Camperdown, New South Wales
  - Research Site, Milton, Queensland
  - Research Site, Melbourne, Victoria
  - Research Site, Perth, Western Australia
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, La Louvière
- Canada (3):
  - Research Site, Newmarket, Ontario
  - Research Site, Lachine, Quebec
  - Research Site, Pointe-Claire, Quebec
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- France (3):
  - Research Site, Lille
  - Research Site, Paris
  - Research Site, Vénissieux
- Germany (3):
  - Research Site, Bad Krozingen
  - Research Site, Dresden
  - Research Site, Heppenheim an der Bergstrasse
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Netherlands (3):
  - Research Site, Alkmaar
  - Research Site, Amsterdam
  - Research Site, Groningen
- Poland (2):
  - Research Site, Lodz
  - Research Site, Warsaw
- South Africa (3):
  - Research Site, Midrand, Gauteng
  - Research Site, Observatory, Western Cape
  - Research Site, Somerset West, Western Cape
- Spain (3):
  - Research Site, Córdoba, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Reus, Catalonia
- Switzerland (2):
  - Research Site, Lugano
  - Research Site, Reinach
- United Kingdom (4):
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Telford
  - Research Site, West Bromwich

REFERENCES:
- [Background] Toth PP, Descamps O, Genest J, Sattar N, Preiss D, Dent R, Djedjos C, Wu Y, Geller M, Uhart M, Somaratne R, Wasserman SM; PROFICIO Investigators. Pooled Safety Analysis of Evolocumab in Over 6000 Patients From Double-Blind and Open-Label Extension Studies. Circulation. 2017 May 9;135(19):1819-1831. doi: 10.1161/CIRCULATIONAHA.116.025233. Epub 2017 Mar 1. PMID 28249876
- [Background] Kuchimanchi M, Grover A, Emery MG, Somaratne R, Wasserman SM, Gibbs JP, Doshi S. Population pharmacokinetics and exposure-response modeling and simulation for evolocumab in healthy volunteers and patients with hypercholesterolemia. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):505-522. doi: 10.1007/s10928-018-9592-y. Epub 2018 May 7. PMID 29736889
- [Background] Cho L, Dent R, Stroes ESG, Stein EA, Sullivan D, Ruzza A, Flower A, Somaratne R, Rosenson RS. Persistent Safety and Efficacy of Evolocumab in Patients with Statin Intolerance: a Subset Analysis of the OSLER Open-Label Extension Studies. Cardiovasc Drugs Ther. 2018 Aug;32(4):365-372. doi: 10.1007/s10557-018-6817-7. PMID 30073585
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Wasserman SM, Sabatine MS, Koren MJ, Giugliano RP, Legg JC, Emery MG, Doshi S, Liu T, Somaratne R, Gibbs JP. Comparison of LDL-C Reduction Using Different Evolocumab Doses and Intervals: Biological Insights and Treatment Implications. J Cardiovasc Pharmacol Ther. 2018 Sep;23(5):423-432. doi: 10.1177/1074248418774043. Epub 2018 May 16. PMID 29768954
- [Background] Cho L, Rocco M, Colquhoun D, Sullivan D, Rosenson RS, Dent R, Xue A, Scott R, Wasserman SM, Stroes E. Design and rationale of the GAUSS-2 study trial: a double-blind, ezetimibe-controlled phase 3 study of the efficacy and tolerability of evolocumab (AMG 145) in subjects with hypercholesterolemia who are intolerant of statin therapy. Clin Cardiol. 2014 Mar;37(3):131-9. doi: 10.1002/clc.22248. Epub 2014 Jan 29. PMID 24477778
- [Background] Stroes E, Colquhoun D, Sullivan D, Civeira F, Rosenson RS, Watts GF, Bruckert E, Cho L, Dent R, Knusel B, Xue A, Scott R, Wasserman SM, Rocco M; GAUSS-2 Investigators. Anti-PCSK9 antibody effectively lowers cholesterol in patients with statin intolerance: the GAUSS-2 randomized, placebo-controlled phase 3 clinical trial of evolocumab. J Am Coll Cardiol. 2014 Jun 17;63(23):2541-2548. doi: 10.1016/j.jacc.2014.03.019. Epub 2014 Mar 30. PMID 24694531
- [Background] Shapiro MD, Minnier J, Tavori H, Kassahun H, Flower A, Somaratne R, Fazio S. Relationship Between Low-Density Lipoprotein Cholesterol and Lipoprotein(a) Lowering in Response to PCSK9 Inhibition With Evolocumab. J Am Heart Assoc. 2019 Feb 19;8(4):e010932. doi: 10.1161/JAHA.118.010932. PMID 30755061
- [Background] Stroes E, Robinson JG, Raal FJ, Dufour R, Sullivan D, Kassahun H, Ma Y, Wasserman SM, Koren MJ. Consistent LDL-C response with evolocumab among patient subgroups in PROFICIO: A pooled analysis of 3146 patients from phase 3 studies. Clin Cardiol. 2018 Oct;41(10):1328-1335. doi: 10.1002/clc.23049. Epub 2018 Oct 21. PMID 30120772
- [Background] Toth PP, Jones SR, Monsalvo ML, Elliott-Davey M, Lopez JAG, Banach M. Effect of Evolocumab on Non-High-Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a): A Pooled Analysis of Phase 2 and Phase 3 Studies. J Am Heart Assoc. 2020 Mar 3;9(5):e014129. doi: 10.1161/JAHA.119.014129. Epub 2020 Mar 2. PMID 32114889
- [Background] Koren MJ, Jones PH, Robinson JG, Sullivan D, Cho L, Hucko T, Lopez JAG, Fleishman AN, Somaratne R, Stroes E. A Comparison of Ezetimibe and Evolocumab for Atherogenic Lipid Reduction in Four Patient Populations: A Pooled Efficacy and Safety Analysis of Three Phase 3 Studies. Cardiol Ther. 2020 Dec;9(2):447-465. doi: 10.1007/s40119-020-00181-8. Epub 2020 Jun 20. PMID 32564340
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women ≥ 18 to ≤ 80 years of age who have tried at least 2 statins and were unable to tolerate any dose or increase in statin dose due to muscle-related side effects were eligible for this study.
  The first participant was enrolled on 24 January 2013 and the last participant enrolled on 29 August 2013.
Pre-assignment Details: Participants received subcutaneous placebo corresponding to the once monthly dose volume during a 6-week screening period. Those who completed the screening period and met final eligibility criteria were randomized 1:1:2:2 into 4 treatment groups. Randomization was stratified by low-density lipoprotein cholesterol (LDL-C) level and statin use.
Period: Overall Study
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Started | 51 | 51 | 103 | 102
Completed | 45 | 50 | 94 | 101
Not Completed | 6 | 1 | 9 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1
Not completed — Decision by sponsor | 5 | 0 | 8 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM | Total
Number analyzed (Participants) | 51 | 51 | 103 | 102 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.1) | 60.2 (8.7) | 60.5 (9.7) | 62.9 (10.2) | 61.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 46 | 46 | 141
  Male | 24 | 29 | 57 | 56 | 166
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 5 | 1 | 10
  Black or African American | 0 | 1 | 3 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  White | 49 | 46 | 94 | 98 | 287
  Other | 1 | 1 | 0 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 2 | 3 | 1 | 7
  Not Hispanic or Latino | 50 | 49 | 100 | 101 | 300
Stratification Factor: Low-density Lipoprotein Cholesterol (LDL-C) Level [Number; unit: participants]
  < 180 mg/dL | 26 | 26 | 52 | 52 | 156
  ≥ 180 mg/dL | 25 | 25 | 51 | 50 | 151
Stratification Factor: Baseline Statin Use [Number; unit: participants]
  No | 41 | 42 | 84 | 82 | 249
  Yes | 10 | 9 | 19 | 20 | 58
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 194.7 (63.8) | 195.2 (51.8) | 192.0 (57.0) | 192.2 (61.2) | 193.1 (58.5)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 231.4 (66.0) | 232.9 (57.0) | 227.9 (56.6) | 222.1 (63.2) | 227.4 (60.4)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 140.0 (37.0) | 140.0 (31.1) | 140.2 (32.1) | 133.1 (32.2) | 137.8 (32.8)
Total Cholesterol/High-Density Lipoprotein Cholesterol Ratio [Mean (Standard Deviation); unit: ratio] | 5.989 (2.190) | 6.137 (1.787) | 5.912 (1.929) | 5.506 (1.925) | 5.827 (1.956)
Apolipoprotein B/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] | 0.943 (0.282) | 1.005 (0.294) | 0.980 (0.318) | 0.901 (0.283) | 0.952 (0.298)
Lipoprotein(a) Concentration [Mean (Standard Deviation); unit: nmol/L] | 106.3 (101.0) | 76.6 (96.7) | 66.2 (72.5) | 70.9 (99.9) | 76.2 (91.9)
Triglyceride Concentration [Mean (Standard Deviation); unit: mg/dL] | 183.4 (79.8) | 187.0 (81.5) | 179.8 (80.0) | 149.3 (63.1) | 171.5 (76.3)
Very Low-density Lipoprotein Cholesterol (VLDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 36.7 (16.0) | 37.1 (15.8) | 35.2 (14.5) | 29.9 (12.6) | 34.0 (14.6)
High-Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 52.4 (18.3) | 48.0 (11.0) | 51.1 (16.4) | 54.0 (16.0) | 51.8 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set (all randomized participants who received at least 1 dose of investigational product (subcutaneously or orally)) with available data (no imputation was performed).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -18.08 (2.52) | -15.05 (2.13) | -56.14 (1.91) | -52.60 (1.58)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; The null hypothesis was that there is no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and ezetimibe, and the alternative hypothesis is that a mean difference does exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model includes treatment group, baseline LDL-C level and statin use, scheduled visit, and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -38.06, 95% CI 2-sided [-43.73 to -32.99], Standard Error of Mean 2.87
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.55, 95% CI 2-sided [-42.16 to -32.94], Standard Error of Mean 2.33

2. Secondary Outcome: Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
mg/dL | -39.1 (5.1) | -33.0 (4.5) | -105.4 (3.9) | -103.6 (3.4)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -66.3, 95% CI 2-sided [-77.9 to -54.7], Standard Error of Mean 5.9
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -70.6, 95% CI 2-sided [-80.5 to -60.7], Standard Error of Mean 5.0

3. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
mg/dL | -36.2 (5.4) | -30.2 (4.7) | -106.0 (4.1) | -99.0 (3.5)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -69.7, 95% CI 2-sided [-82.0 to -57.5], Standard Error of Mean 6.2
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.8, 95% CI 2-sided [-79.2 to -58.4], Standard Error of Mean 5.3

4. Secondary Outcome: Percentage of Participants With Mean LDL-C at Weeks 10 and 12 of Less Than 70 mg/dL (1.8 mmol/L)
Time Frame: Weeks 10 and 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percentage of participants | 2.0 [0.4 to 10.5] | 0.0 [0.0 to 7.3] | 45.5 [36.2 to 55.2] | 42.0 [32.8 to 51.8]
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by baseline LDL-C and statin use. For testing, non-achievement was imputed for participants with missing data; Treatment Difference = 43.5, 95% CI 2-sided [30.9 to 53.4]
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 4, analysis 1]; Treatment Difference = 42.0, 95% CI 2-sided [30.3 to 51.8]

5. Secondary Outcome: Percentage of Participants With LDL-C < 70 mg/dL (1.8 mmol/L) at Week 12
Time Frame: Week 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percentage of participants | 2.0 [0.4 to 10.7] | 0.0 [0.0 to 7.9] | 50.0 [40.3 to 59.7] | 37.5 [28.5 to 47.5]
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 4, analysis 1]; Treatment Difference = 48.0, 95% CI 2-sided [35.0 to 57.8]
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 4, analysis 1]; Treatment Difference = 37.5, 95% CI 2-sided [25.5 to 47.5]

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -17.18 (2.15) | -14.54 (1.86) | -48.72 (1.64) | -49.13 (1.40)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.53, 95% CI 2-sided [-36.34 to -26.73], Standard Error of Mean 2.43
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.58, 95% CI 2-sided [-38.63 to -30.54], Standard Error of Mean 2.05

7. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -16.53 (2.30) | -13.16 (1.93) | -48.62 (1.74) | -46.15 (1.43)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.09, 95% CI 2-sided [-37.28 to -26.90], Standard Error of Mean 2.63
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.99, 95% CI 2-sided [-37.19 to -28.79], Standard Error of Mean 2.12

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full anlaysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -13.67 (2.15) | -11.02 (2.21) | -45.88 (1.68) | -46.01 (1.65)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.20, 95% CI 2-sided [-36.92 to -27.49], Standard Error of Mean 2.39
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.99, 95% CI 2-sided [-39.59 to -30.39], Standard Error of Mean 2.33

9. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -12.95 (2.32) | -9.97 (2.34) | -45.81 (1.79) | -43.07 (1.73)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.86, 95% CI 2-sided [-38.04 to -27.68], Standard Error of Mean 2.62
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.10, 95% CI 2-sided [-38.04 to -28.17], Standard Error of Mean 2.50

10. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/High Density Lipoprotein Cholesterol Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -13.44 (2.14) | -11.20 (2.16) | -40.83 (1.65) | -41.14 (1.62)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.39, 95% CI 2-sided [-32.11 to -22.67], Standard Error of Mean 2.39
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -29.94, 95% CI 2-sided [-34.72 to -25.17], Standard Error of Mean 2.42

11. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/High Density Lipoprotein Cholesterol Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -14.13 (2.30) | -9.92 (2.34) | -40.42 (1.75) | -38.57 (1.73)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -26.28, 95% CI 2-sided [-31.42 to -21.15], Standard Error of Mean 2.60
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.66, 95% CI 2-sided [-33.88 to -23.43], Standard Error of Mean 2.64

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -13.00 (2.27) | -11.94 (2.56) | -47.86 (1.77) | -48.31 (1.92)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.86, 95% CI 2-sided [-39.84 to -29.88], Standard Error of Mean 2.52
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.37, 95% CI 2-sided [-41.73 to -31.01], Standard Error of Mean 2.71

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -13.14 (2.47) | -11.37 (2.71) | -47.66 (1.90) | -45.51 (2.01)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.53, 95% CI 2-sided [-40.05 to -29.00], Standard Error of Mean 2.79
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.13, 95% CI 2-sided [-39.87 to -28.39], Standard Error of Mean 2.91

14. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -2.30 (3.36) | 1.55 (4.01) | -26.20 (2.64) | -23.72 (2.97)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -23.90, 95% CI 2-sided [-31.27 to -16.54], Standard Error of Mean 3.73
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.26, 95% CI 2-sided [-33.75 to -16.77], Standard Error of Mean 4.30

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -1.74 (3.58) | 5.81 (5.10) | -27.03 (2.78) | -22.07 (3.66)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.29, 95% CI 2-sided [-33.26 to -17.33], Standard Error of Mean 4.03
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.88, 95% CI 2-sided [-39.21 to -16.56], Standard Error of Mean 5.73

16. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -3.74 (3.88) | -0.32 (4.65) | -6.32 (2.94) | -6.73 (3.44)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.97, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -2.59, 95% CI 2-sided [-11.38 to 6.20], Standard Error of Mean 4.45
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.33, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -6.42, 95% CI 2-sided [-16.55 to 3.71], Standard Error of Mean 5.13

17. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -5.47 (4.25) | 2.16 (5.52) | -3.88 (3.18) | -2.53 (3.98)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.97, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 1.58, 95% CI 2-sided [-8.14 to 11.31], Standard Error of Mean 4.92
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.33, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -4.69, 95% CI 2-sided [-17.04 to 7.67], Standard Error of Mean 6.25

18. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | 0.33 (1.98) | 1.44 (2.03) | 5.48 (1.51) | 7.18 (1.51)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.068, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 5.15, 95% CI 2-sided [0.74 to 9.56], Standard Error of Mean 2.23
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.13, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 5.74, 95% CI 2-sided [1.23 to 10.24], Standard Error of Mean 2.28

19. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | 1.77 (2.22) | 1.64 (2.22) | 5.34 (1.67) | 6.47 (1.63)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.068, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 3.57, 95% CI 2-sided [-1.49 to 8.63], Standard Error of Mean 2.56
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.13, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 4.83, 95% CI 2-sided [-0.16 to 9.81], Standard Error of Mean 2.52

20. Secondary Outcome: Percent Change From Baseline in Very Low-Density Lipoprotein Cholesterol at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -5.76 (3.80) | -2.93 (4.41) | -7.60 (2.89) | -6.46 (3.21)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.97, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -1.84, 95% CI 2-sided [-10.43 to 6.75], Standard Error of Mean 4.35
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.33, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -3.53, 95% CI 2-sided [-13.12 to 6.06], Standard Error of Mean 4.85

21. Secondary Outcome: Percent Change From Baseline in Very Low-Density Lipoprotein Cholesterol at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -5.49 (4.05) | -2.25 (5.11) | -6.16 (3.08) | -2.18 (3.60)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.97, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -0.67, 95% CI 2-sided [-9.96 to 8.61], Standard Error of Mean 4.70
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.33, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 0.08, 95% CI 2-sided [-11.24 to 11.39], Standard Error of Mean 5.72

22. Primary Outcome: Percent Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set with available data (no imputation was performed).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 51 | 51 | 103 | 102
percent change | -19.21 (2.40) | -16.62 (2.03) | -56.11 (1.83) | -55.31 (1.53)
Statistical Analysis 1: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; The null hypothesis was that there is no mean difference in the percent change from Baseline in the average value of LDL-C at Weeks 10 and 12 between evolocumab and ezetimibe, and the alternative hypothesis is that a mean difference does exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.90, 95% CI 2-sided [-42.26 to -31.55], Standard Error of Mean 2.71
Statistical Analysis 2: Comparison: Ezetimibe (QM) vs Evolocumab QM; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -38.69, 95% CI 2-sided [-43.06 to -34.22], Standard Error of Mean 2.21

ADVERSE EVENTS:
Time Frame: From the first dose of blinded investigational product until the end of the study (up to 14 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Serious Adverse Events (participants affected / at risk) | 1/51 | 3/51 | 5/103 | 1/102
Other Adverse Events (participants affected / at risk) | 20/51 | 29/51 | 28/103 | 42/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ezetimibe (Q2W) (N=51) | Ezetimibe (QM) (N=51) | Evolocumab Q2W (N=103) | Evolocumab QM (N=102)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cartilage graft (Surgical and medical procedures) | 0 | 0 | 0 | 1
Osteotomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Spinal decompression (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ezetimibe (Q2W) (N=51) | Ezetimibe (QM) (N=51) | Evolocumab Q2W (N=103) | Evolocumab QM (N=102)
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 5 | 3 | 6
Fatigue (General disorders) | 4 | 6 | 3 | 6
Injection site erythema (General disorders) | 0 | 3 | 2 | 2
Influenza (Infections and infestations) | 3 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 5 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 11 | 7 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 12
Headache (Nervous system disorders) | 3 | 6 | 4 | 12
Paraesthesia (Nervous system disorders) | 1 | 4 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.